CLINICAL TRIAL: NCT02905305
Title: Pilot Evaluation of Combined Investigational Device: CI4CID With Controlled Dosage of Dexamethasone
Brief Title: Cochlear Implant With Anti-Inflammatory Agent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hearing Cooperative Research Centre (Other)
Collaborators: Cochlear (Industry); Royal Victoria Eye and Ear Hospital (Other Government); Royal Prince Alfred Hospital, Sydney, Australia (Other); St Vincent's Hospital Melbourne (Other); Westmead Hospital, New South Wales (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLTD 5495
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Hearing Loss
Keywords: cochlear implants; Dexamethasone; combined device
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CA with dexamethasone base (Experimental): Contour Advance electrode with controlled dose of dexamethasone base
  Interventions: Device: Contour Advance electrode with controlled dose of dexamethasone base
- Contour Advance (Active Comparator): Standard Contour Advance electrode array
  Interventions: Device: Contour Advance electrode

INTERVENTIONS:
Device: Contour Advance electrode with controlled dose of dexamethasone base — The Combined Device consists of a standard cochlear implant receiver-stimulator coupled to a Contour Advance electrode loaded with a controlled dose of dexamethasone base.
  Arms: CA with dexamethasone base
Device: Contour Advance electrode — Standard Contour Advance electrode
  Arms: Contour Advance

SUMMARY:
In an effort to further preserve residual acoustic hearing after cochlear implantation, it may be beneficial to incorporate anti-inflammatory agents into the electrode array for passive elution over a time course after implantation. This study aims to assess the ease and effectiveness of such an electrode design, and to assess the preliminary safety of use of such a device in the post-operative period. This study is a first-time-in-human study of the investigational device.

In the first instance, the aim of the current investigation is to obtain first experience in use of a Combined Device in the adult clinical population, and to assess tools and techniques that may be considered in future clinical studies of similar devices.

ELIGIBILITY:
Inclusion Criteria:

1. Duration severe to profound hearing impairment in implanted ear of less than or equal to 30 years
2. Post-lingual hearing impairment defined as onset of hearing loss at greater than two years of age
3. Evidence of Pneumovax vaccination within three years of implantation date (for subjects to be implanted with the investigational device)

Exclusion Criteria:

1. Ossification or any other cochlear anomaly that might prevent complete insertion of the electrode array or increased risk of infection (i.e. dysplastic cochlea), as confirmed by medical examination and imaging including MRI
2. Current use of grommets or evidence of tympanic membrane perforation
3. Known allergic reaction to dexamethasone or similar medicine
4. Diagnosis of Auditory Neuropathy
5. Active middle ear infection or history of middle ear infection within past two years
6. Unrealistic expectations on the part of the subject regarding the possible benefits, risks, and limitations that are inherent to the surgical procedure and use of the prosthetic device
7. Unwillingness or inability of the candidate to comply with all investigational requirements
8. Additional disabilities that would prevent or restrict participation in the audiological and medical evaluations required of the clinical investigation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-09-10 (Actual); Primary Completion 2017-11-06 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Surgical feedback | During surgery
  Questionnaire used to obtain surgical feedback from experienced cochlear implant surgeons regarding the electrode design, and ease and effectiveness of surgery, when using the Combined Device as compared to the Contour Advance electrode
Safety of Combined Device | Monitoring over 24 months
  Monitoring of device related adverse events that occur during the study period, to assess the preliminary safety of the Combined Device

SECONDARY OUTCOMES:
Electrode impedance | Testing over 24 months
Electrically evoked compound action potential (ECAP) | Testing over 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- The HEARing CRC, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No